CLINICAL TRIAL: NCT03839719
Title: Efficacy of Ocimum Sanctum as a Pre-procedural Mouth Rinse in Reducing Aerosol Contamination Produced by Ultrasonic Scaler: a Clinical and Microbiological Study.
Brief Title: OSE as a Pre-procedural Mouth Rinse: A Clinical and Microbiological Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Dr. Pratik kumar Ashok bhai Chaudhari, Principal Investigator, Government College of Dentistry, Indore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 052/IEC/SS/2019
Record Dates: First submitted 2019-02-01; First posted 2019-02-15 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Gingivitis; Periodontitis; Aerosol Disease; Gingival Disease; Periodontal Diseases
Keywords: Gingivitis; Aerosol; Ocimum sanctum; Mouth rinse; SRP; Chlorhexidine mouthrinse; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis; Gingival Diseases; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Ultrasonic scaling was done in the 1st and 4th quadrant without any mouth rinse and fall out samples were collected in the blood agar plates kept at a distance of 0.5 m and 1 m from the oral cavity. After ultrasonic scaling of the 1st and 4th quadrant minimum 30min interval maintained. After interval of 30min rinsing the mouth with the either OC/CHX/Placebo (OC= Ocimum sanctum mouthrinse, CHX=Chlorhexidine Gluconate mouthrinse) mouthrinse) done for 60s, Ultrasonic scaling was again done in the 2nd and 3rd quadrant and fall out samples were collected in the newly placed blood agar plates kept at 0.5 m and 1 m away from the patient. Treatment was carried out by placing 03 sterile agar plates uncovered at pre-designated sites to collect samples of aerosolized bacteria After ultrasonic scaling of the 1st and 4th quadrant and after 2nd and 3rd quadrant.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This single-center, double-masked, placebo-controlled study was conducted over a period of 02 months. The participants and investigator are blinded about mouthrinse use and assigned quadrant.
  Then Ultrasonic scaling was done in the 1st and 4th quadrant without any mouth rinse and Ultrasonic scaling is done in the 2nd and 3rd quadrant by giving either OC/CHX/Placebo mouth rinse
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group OC (Experimental): Ocimum sanctum (OC) is a natural herb which is known for its broad spectrum medicinal properties. Ocimum sanctum is also listed by the U.S. FDA as an herb Generally Recognized As Safe (GRAS) for its intended use as a therapeutic herb. Pharmacological constitutes present in the extract are eugenol, Urosolic acid, Carvacrol, linalool , limatrol, caryophyllene, and methyl carvicol. The literature showed that Ocimum sanctum extract has significant anti-gingivitis and anti-inflammatory effect as mouthrinse.
  Other Names:
  Tulsi Holy Basil
  Interventions: Procedure: Group OC; Procedure: Group CHX
- Group CHX (Active Comparator): Chlorhexidine Gluconate (C34H54Cl2N10O14) is a bisbiguanide formulation with cationic properties. A literature review, highlighting chlorhexidine as not only a plaque control agent but also as an effective antimicrobial agent and its wider application in a variety of oral disorders in various formulations.
  As an antimicrobial agent, chlorhexidine is effective in vitro against both Gram-positive and Gram-negative bacteria including aerobes and anaerobes and yeasts and fungi. The digluconate of chlorhexidine (1:6Di 4' chlorophenyl-diguani-dohexane) is a synthetic antimicrobial drug which has been widely used as a broad spectrum antiseptic.
  Other Names:
  Chlorhexidine
  Interventions: Procedure: Group OC; Procedure: Group CHX
- Group PI (Placebo Comparator): Group PI: Placebo (Distilled water) as the mouthrinse.
  Placebo (Distilled water) 10 ml is used as mouthrinse. Distilled water is commonly used as an excipient in a variety of drugs and it is also widely used as a placebo.
  Ultrasonic scaling was done in the 1st and 4th quadrant without any mouth rinse (placebo mouthrinse) and fall out samples were collected in the blood agar plates kept at a distance of 0.5 m and 1 m from the oral cavity.
  Treatment was carried out by placing 03 sterile agar plates uncovered at pre-designated sites to collect samples of aerosolized bacteria.
  Interventions: Procedure: Group PI

INTERVENTIONS:
Procedure: Group PI — Before rinsing with the mouthrinse, Ultrasonic scaling was done in the 1st and 4th quadrant without any mouth rinse (placebo mouthrinse) and fall out samples were collected in the blood agar plates kept at a distance of 0.5 m and 1 m from the oral cavity.
  Other Names: mouthrinse followed by Ultrasonic scaling
  Arms: Group PI
Procedure: Group OC — After ultrasonic scaling of the 1st and 4th quadrant minimum 30min interval maintained. After interval of 30min rinsing the mouth with the either OC/CHX/Placebo (OC= Ocimum sanctum mouthrinse, CHX=Chlorhexidine Gluconate mouthrinse) mouthrinse) done for 60s, Ultrasonic scaling was again done in the 2nd and 3rd quadrant and fall out samples were collected in the newly placed blood agar plates kept at 0.5 m and 1 m away from the patient.
  Other Names: mouthrinse followed by Ultrasonic scaling
  Arms: Group CHX; Group OC
Procedure: Group CHX — After ultrasonic scaling of the 1st and 4th quadrant minimum 30min interval maintained. After interval of 30min rinsing the mouth with the either OC/CHX/Placebo (OC= Ocimum sanctum mouthrinse, CHX=Chlorhexidine Gluconate mouthrinse) mouthrinse) done for 60s, Ultrasonic scaling was again done in the 2nd and 3rd quadrant and fall out samples were collected in the newly placed blood agar plates kept at 0.5 m and 1 m away from the patient.
  Other Names: Mouthrinse followed by Ultrasonic scaling
  Arms: Group CHX; Group OC

SUMMARY:
* Periodontal disease- Inflammatory, Multifactorial, and Threshold disease. Periodontal disease is a highly prevalent dental disease, an almost 100% prevalence in developing countries.
* Non-surgical periodontal includes scaling and root planing (SRP) an essential part of successful periodontal therapy.
* The spread of infection through aerosol and splatter has long been considered one of the main reason for the possible transmission of infectious agents and their ill effects on The Health of patients and Dental Health care Professionals.
* Aerosols are generated during Tooth preparation/Rotary instrument/ air abrasion/Air-water syringe, Ultrasonic scaler, and while doing Air polishing.
* Studies have also reported an association of these aerosols with Respiratory infections, Ophthalmic and Skin infections, Tuberculosis, and Hepatitis B. current research suggests that having patients use an antimicrobial rinse before treatment may decrease microbial aerosols.
* Chlorhexidine mouthwash is regarded as Gold Standard mouthwash but, have many local side effects including have many local side effects including extrinsic tooth and tongue brown staining, taste disturbance, enhanced supragingival calculus formation, less commonly, desquamation of oral mucosa, and even liver damage in rats.
* In the emerging era of pharmaceuticals, herbal medicines with their naturally occurring active ingredients offer a gentle and enduring way for the restoration of health by the least harmful method.
* Ocimum Sanctum (Tulsi) is known as THE QUEEN OF HERBS effective in reducing plaque accumulation, gingival inflammation, and bleeding & has no side effects as compared to Chlorhexidine. Very few studies which can be counted on fingers have been conducted worldwide in this direction, globally showing their beneficial effects.

DETAILED DESCRIPTION:
The spread of infection through aerosol and splatter has long been considered one of the main reason for the possible transmission of infectious agents and their ill effects on the health of patients and dental health care professionals. Aerosol and splatter are a concern in dentistry because of their potential effects on the health of immuno-compromised patients and of dental personnel. These aerosols may be inhaled into the lungs to reach the alveoli or may come in contact with the skin or mucous membranes. Most of the aerosols produced during treatment procedures have a diameter of 5μm or less, and these can cause respiratory or other health problems because they can penetrate into, and remain within the lungs. The oral cavity consists of billions and billions of microorganisms, which can get transmitted from one person to another through water contamination, surface contact or through aerosols. Aerosols are generated during tooth preparation with a rotary instrument or air abrasion, during the use of an air-water syringe, ultrasonic scaler, and while doing air polishing. Miller (1976) found that aerosols generated from patients' mouths contained up to a million bacteria per cubic foot of air.

All health care professionals including the dentists, dental hygienists, and nurses can get exposed to microorganisms present in patients' blood, saliva and from instruments, which can lead to cross infections. The oral cavity harbors numerous bacteria and viruses from the respiratory tract, dental plaque, and oral fluids. Viruses which are present in aerosols such as human immunodeficiency virus hepatitis B can penetrate the conjunctiva, respiratory tract of clinician, assistant, and patients. In addition to this, some viruses such as mumps, rubella, and influenza also pose a serious risk to health care professionals. Any dental procedure that has the potential to aerosolize saliva will cause contamination of air with organisms from some or all of these sources. Other studies have also reported an association of these aerosols with respiratory infections, ophthalmic and skin infections, tuberculosis, and hepatitis B. Current research suggests that having patients use an antimicrobial rinse before treatment may decrease microbial aerosols.

Chlorhexidine gluconate, a bisbiguanide, is considered to be the gold standard of antimicrobial rinses because of broad-spectrum antibacterial activity but, it also has some side effects, notably tooth staining, taste alteration, enhanced supragingival calculus formation and less commonly desquamation of the oral mucosa. Also other then Chlorhexidine Providone iodine and essential oils are commonly used as mouthrinse.

In the emerging era of pharmaceuticals, herbal medicines with their naturally occurring active ingredients offer a gentle and enduring way for the restoration of health by the least harmful method. Herbal medicine is both promotive and preventive in its approach. Also, herbal mouth rinses with their natural ingredients offer a safe and effective option as mouthrinse.

The herbal mouthwash used in this study is made from natural herb extracts of Ocimum sanctum. Ocimum sanctum is commonly known as 'Tulsi' and popularly known as 'The Queen of Herbs', and the "Mother Medicine of Nature" due to its perceived medicinal qualities. Tulsi extract has been widely used in traditional medicine and human clinical trial without significant side effects. Scientific investigations during the last several decades have shown that various parts of Ocimum sanctum, including leaves, stem, root, flowers, and seed, have a plethora of biological and pharmacological activities, including antioxidant, anti-inflammatory, antiallergic, immunomodulatory, antimicrobial etc.

Looking into the above background, The investigators hypothesized the beneficial effects of Pre-procedural rinsing with an antimicrobial mouthrinse in reducing the level of viable bacteria contained in aerosols generated by ultrasonic scaling. Also, very few studies are conducted on herbal products as a pre-procedural mouthrinse therefore, the study should be conducted to gain evidence regarding their effectiveness. So, The investigators have planned to conduct this study.

This study has been planned and would be conducted in the Department of Periodontology, Govt. College of Dentistry, Indore (M.P.). A minimum of 60 Recruited Outdoor Patients age group of 18-40 years, who abide by approved protocol guidelines, and are ready to give written informed consent are enrolled for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Cases with Generalized Chronic Gingivitis or cases with mild
2. Generalized Chronic Periodontitis patients of any sex.
3. Systemically healthy individuals.
4. Patient having ≥ 20 teeth.
5. Patients in the age group of 18-40 years, who abide by approved protocol guidelines, and are ready to give written informed consent.

Exclusion Criteria:

1. Any known systemic disease which has effects on periodontium such as diabetes, cardiovascular, cancer etc.
2. Patients on anti-inflammatory, perioceutics, antibiotics, steroids, cytotoxic and drugs since 03 months.
3. Patients who have known allergy to the material used for the study.
4. Pregnant and lactating mothers.
5. Patients had undergone any kind of nonsurgical and/or surgical periodontal therapy earlier, in the past 6 months.
6. Tobacco users (smoke and smokeless) and alcoholics.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Counting of the colony-forming units (CFU) | Up to 48 hr
  Preformed 10% blood agar plates were used which were incubated at 37°C for 48 hr after collecting the sample. Counting of the colony-forming units (CFU) was performed by the microbiologist, who was blinded regarding the time of exposure and location of agar plate. The microbial counting was done after that.

CONTACTS AND LOCATIONS:
Overall Officials: DR.MADHU S. RATRE, M.D.S., Study Director — Govt. college of dentistry, Indore
Locations (1):
- Department of periodontology, GDC Indore, Indore, Madhu Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gupta G, Mitra D, Ashok KP, Gupta A, Soni S, Ahmed S, Arya A. Efficacy of preprocedural mouth rinsing in reducing aerosol contamination produced by ultrasonic scaler: a pilot study. J Periodontol. 2014 Apr;85(4):562-8. doi: 10.1902/jop.2013.120616. Epub 2013 Jul 15. PMID 23855840
- [Result] Reddy S, Prasad MG, Kaul S, Satish K, Kakarala S, Bhowmik N. Efficacy of 0.2% tempered chlorhexidine as a pre-procedural mouth rinse: A clinical study. J Indian Soc Periodontol. 2012 Apr;16(2):213-7. doi: 10.4103/0972-124X.99264. PMID 23055587
- See also: Efficacy of preprocedural mouth rinsing in reducing aerosol contamination produced by ultrasonic scaler: a pilot study. — https://www.ncbi.nlm.nih.gov/pubmed/23855840
- See also: Efficacy of 0.2% tempered chlorhexidine as a pre-procedural mouth rinse: A clinical study. — https://www.ncbi.nlm.nih.gov/pubmed/23055587